CLINICAL TRIAL: NCT05569187
Title: An Observational, Retrospective, Multicenter, National Study of the Effectiveness of Ribociclib in Combination With Non-steroidal Aromatase Inhibitors in First-line Treatment of Brazilian Patients With HR+/HER2- Advanced Breast Cancer
Brief Title: Ribociclib in Combination With Non-steroidal Aromatase Inhibitors in Patients With Advanced Breast Cancer
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLEE011ABR02
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer
Keywords: HR+/HER2-,; advanced breast cancer,; ribociclib,; non-steroidal aromatase inhibitors,; first-line treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Ribociclib in combination with non-steroidal aromatase inhibitors: Included patients who received doses (600 mg, 400 mg, and 200 mg) at 6 months and 1 year
  Interventions: Drug: Ribociclib

INTERVENTIONS:
Drug: Ribociclib — Included patients who received doses (600 mg, 400 mg, and 200 mg) at 6 months and 1 year

SUMMARY:
Observational, longitudinal (retrospective cohort), multicenter, national study aiming to evaluate the proportion of women with HR+/HER2- advanced breast cancer treated with ribociclib plus non-steroidal aromatase inhibitors who were alive and without disease progression at 1 year.

DETAILED DESCRIPTION:
The study was conducted in 11 Brazilian sites specialized in the treatment of this condition. The study data were collected from the review of medical records by the Investigator (or designated).

The sites must have had adequate medical records to ensure robust medical record review. Therefore, a feasibility assessment was carried out at potential site prior to the study implementation to assess the adequacy of medical records and the data routinely available.

ELIGIBILITY:
Inclusion criteria

* Female patient ≥ 18 years of age. All the patients must have at least one year of follow-up
* Patients at an age not consistent with postmenopausal status could only participate if they had oophorectomy surgery or being on treatment with goserelin for ovarian suppression Post-menopausal women defined as age ≥ 60 years old or < 60 years old and amenorrhea for 12 months or more (in the absence of chemotherapy, tamoxifen, toremifene or goserelin use for ovarian suppression)
* Confirmed diagnosis of HR+/HER2- locally advanced or metastatic BC
* Never in use of CDK 4/6i

Exclusion criteria

* Patients in menopause status other than postmenopausal (young patients must have undergone oophorectomy being on treatment with goserelin for ovarian suppression to be characterized as postmenopausal)
* Previous use, at any time, of CDK 4/6i
* The patient received any previous systemic therapy for advanced breast cancer Patients who have received (neo)adjuvant therapy for breast cancer are eligible. If previous (neo) adjuvant therapy has included letrozole or anastrozole, the disease- free interval should be longer than 12 months from completion of treatment until entry in this trial Patients who received ≤28 days of letrozole or anastrozole for advanced disease prior to inclusion in this trial are eligible
* Uncontrolled heart disease and/or clinically significant cardiac repolarization abnormalities

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study included women with HR+/HER2- advanced breast cancer treated with ribociclib plus non-steroidal aromatase inhibitors
Study Population: The study population was composed only of women aged 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Proportion of patients alive and progression-free from disease at 1 year | 1 year post-treatment
  The purpose was to evaluate the effectiveness of first-line ribociclib in combination with non-steroidal aromatase inhibitors in a Brazilian female population diagnosed with HR+/HER2- locally advanced or metastatic BC. Effectiveness was measured by the proportion of patients alive and free of disease progression at 1 year.

SECONDARY OUTCOMES:
Proportion of patients alive and progression-free from disease at 6 months | 6 months post-treatment
  The purpose was to evaluate the effectiveness of first-line ribociclib in combination with non-steroidal aromatase inhibitors in a Brazilian female population diagnosed with HR+/HER2- locally advanced or metastatic BC. Effectiveness was measured by the proportion of patients alive and free of disease progression at 6 months post-treatment.
Proportion of patients who had disease progression at 6 months | 6 months post-treatment
  The purpose was to evaluate the proportion of patients who had disease progression at 6 months.
Proportion of patients who had disease progression at 1 year | 1 year post-treatment
  The purpose was to evaluate the proportion of patients who had disease progression at 1 year.
Proportion of patients who died at 6 months | 6 months post-treatment
  The purpose was to evaluate the proportion of patients who died at 6 months.
Proportion of patients who died at 1 year | 1 year post-treatment
  The purpose was to evaluate the proportion of patients who died at 1 year.
Proportion and cause of patients who reduced a treatment dose at 6 months | 6 months post-treatment
  Patients who reduced a treatment dose (from 600 mg to 400 mg or from 400 mg to 200 mg)
Proportion and cause of patients who reduced a treatment dose at 1 year | 1 year post-treatment
  Patients who reduced a treatment dose (from 600 mg to 400 mg or from 400 mg to 200 mg)
Frequency of dose interruption and cause, per patient, at 1 year | 1 year post-treatment
  The purpose was to evaluate frequency of dose interruption and cause, per patient, at 1 year.
Adverse Event frequency and classification of the severity degree | throughout the study, approximately 1 year
  Frequency and classification of the degree of severity of the following adverse events of interest: neutropenia, febrile neutropenia, increased QT interval (> 60 ms,> 480ms ≤ 500 ms, and> 500 ms), AST/ALT elevation three times greater than upper limit. In relation to the adverse events of interest, they were classified regarding the severity, graded from 1 to 4, corresponding to mild, moderate, severe and life-threatening, or as described in the medical record.
Pattern of the treatment of AE of interest at 6 months | 6 months post-treatment
  Pattern of the treatment of AE of interest were reported to evaluate how the patients with AE of interest were treated.
Pattern of the treatment of AE of interest at 12 months | 12 months post-treatment
  Pattern of the treatment of AE of interest were reported to evaluate how the patients with AE of interest were treated.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CLEE011ABR02 from the Novartis Clinical Trials Website — http://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17980